CLINICAL TRIAL: NCT07143058
Title: Flaps of Head and Neck in Oral Cancer
Brief Title: Different Modalities Flaps of Head and Neck Reconstructions in Oral Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Ahmed Mohamed Abdelhafiz (Other)
Collaborators: Sohag University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Abdelhafiz, Resident in general surgery department, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-25-6__15MS
Record Dates: First submitted 2025-06-29; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Oral Cancer
Keywords: Different Modalities of Flaps used in Head and Neck Reconstructions in oral cancer Patients, retrospective study
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Flaps reconstruction in head and neck in oral cance — Follow up and quality of life of reconstruction flaps in head and neck
Procedure: Flap of head and neck — All types of flaps in oral cancer reconstruction

SUMMARY:
Different Modalities of Flaps used in Head and Neck Reconstructions in oral cancer Patients, retrospective study

Study design:

This study will be conducted in a Retrospective study with prospective collective data. At General Surgery Department of Sohag University Hospital in the period between June 2020 to June 2025. Data base will be gathered, reviewed, and consequently will be analyzed.

Study population:

The study will include patients presented post operative Head and Neck cancer Resection and Reconstruction with flap during the period of the study, analysis of the clinical presentation, follow up size, color, regeneration skin, early and late complication and a defect appear

Inclusion criteria:

All patients with head and neck Reconstruction on oral cancer patients

1. Age: any age.
2. Sex: males and females.
3. Cooperative, mentally healthy.

Exclusion criteria :

Patients with associated with

1 -Severe chronic illness such as chronic renal failure, chronic liver disease, etc.

2- Mentally or psychologically disordered patients.

DETAILED DESCRIPTION:
Follow up:

The following diameters of patients will be entered into a dedicated database:

Quality of life Questionnaire survey Washington University

2- Clinical: Age. Gender. Comorbidity disease Type , size and site of Tumor Pathology of Tumor Resected part and Method of Resection Size and color of flap Cosmeses Early and late complication Revision of Reconstruction 3 -Investigation: Lab Cbc, Esr, Crp, d-dimer

Radiological:

Ultrasonography laser intervention Statistical method of study Statistical analysis will be done by SPSS v26 (IBM Inc., Chicago, IL, USA). Shapiro-Wilks test and histograms will be used to evaluate the normality of the distribution of data. Quantitative parametric data will be presented as mean and standard deviation (SD). Quantitative non-parametric data will be presented as median and interquartile range (IQR). Qualitative variables will be presented as frequency (%).

Ethical consideration:

Anoralandwrittenconsent willbetakenfromthepatientsincludedinthestudyand willbeintroducedtoethicsscientificcommitteeatSohagUniversityhospitalforapproval.

ELIGIBILITY:
Inclusion Criteria :

All patients with head and neck Reconstruction on oral cancer patients ,Cooperative and mentally healthy

Exclusion Criteria:Patients with associated with Severe chronic illness such as chronic renal failure, chronic liver disease, etc.

Mentally or psychologically disordered patients

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with oral cancer done flap reconstruction
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | Up to 1 week
  how many days staying in hospital post sugery of reconstrucion of head and neck
incidence of infection | Up to 1 week
  incidence of wound infection , discharge pus ,edema ,how many days to releved by antibiotic
incidence of Bleeding | Up to 1 week
  incidence of bleeding and hematoma under flap which cause compromise of local flap vascularity by inducing vasospasm, stretching the sub dermal plexus, or separating the flap from the surface of the recipient site
incidence of Ischemia | Up to 1 week
  incidence of ischemia of flap as dark skin , Pale, cold, delayed capillary refill, no bleeding on needle prick.
Wound Dehiscence | Up to 4 weeks
  : The surgical wound may separate, exposing the flap
Fistula Formation | Up to 4 weeks
  An abnormal connection can form between the flap and other structures, like the oral cavity or pharynx , clinically leakage and ct neck e iv contrast or mri show track of fistula
Number of participants with fibrosis | Up to 8 weeks
  may occur fibrosis between flap and beside structures of oral cavity ,make limitation of movement of mandible , mri image show fibrosis
questionnaire quality of life of Washington university : Health-related quality of life (HRQOL) is an important outcome parameter following treatment for head and neck cancer. | 1 year after surgery
  . Version 4 of the UW-QOL questionnaire consists of 12 single question domains, these having between 3 and 6 response options that are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response. The domains are pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood and anxiety. Another question asks patients to choose up to three of these domains that have been the most important to them.There are also three global questions, one about how patients feel relative to before they developed their cancer, one about their health-related QOL and one about their overall QOL..Scoring of UW-QOL domains The UW-QOL has domains based upon discrete ordinal responses. Scoring is scaled to so that a score of 0 represents the worst possible response, and a score of 100 represents the best possible response .http://www.hancsupport.com/professionals/quality-life/qol-questionnaires/uw-hrqol/uw-qol-v4-translations

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university faculty of medicine, Sohag, Egypt